CLINICAL TRIAL: NCT03494192
Title: Utilizing Scapula Retraction Exercises With or Without Glenohumeral Rotational Exercises With a Gradual Progression: A Double-Blind Randomized Controlled Trial for Subacromial Pain Syndrome
Brief Title: Effects of Exercise Trainings on Pain, Function and AHD in Patients With SPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Leyla Eraslan, PhD Candidate, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA-180018
Record Dates: First submitted 2018-03-27; First posted 2018-04-11 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Subacromial Impingement Syndrome
Keywords: acromiohumeral distance; pain; functional level; Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- scapula retraction exercise group (Experimental): * Manual Therapy
  * Stretching Exercises
  * Exercise training focus on scapulothoracic muscles will be applied two times per week total 12 week After 12 week follow-up, patients will proceed to reduced exercise program until the 6-month follow-up.
  Interventions: Other: Scapula Retraction Exercise Group
- Scapula Retraction +Glenohumeral Rotational Exercise Group (Experimental): * Manual Therapy
  * Stretching Exercises
  * Exercise training focus on scapulothoracic muscles
  * Exercise training focus on rotator cuff muscles will be applied two times per week total 12 week After 12 week follow-up, patients will proceed to reduced exercise program until the 6-month follow-up.
  Interventions: Other: Scapula Retraction +Glenohumeral Rotational Exercise Group
- Control Group (No Intervention): Age-sex and hand-dominancy matched healthy controls will be included as a control group (CG) for acromiohumeral distance (AHD) normative data

INTERVENTIONS:
Other: Scapula Retraction Exercise Group — physiotherapy program consists of manual therapy, supervised stretching and scapulothoracic muscles strengthening exercises and home exercise programme including stretching and strengthening exercises will be applied two times a week total 24 sessions.
  After 24 sessions completed, patients will proceed to reduced exercise program until the 6-month follow-up.
  Other Names: scapula stabilization exercises
  Arms: scapula retraction exercise group
Other: Scapula Retraction +Glenohumeral Rotational Exercise Group — physiotherapy program consists of manual therapy, supervised stretching and scapulothoracic and also rotator cuff muscles strengthening exercises and home exercise programme including stretching and strengthening exercises will be applied two times a week total 24 sessions.
  After 24 sessions completed, patients will proceed to reduced exercise program until the 6-month follow-up
  Other Names: Scapula stabilization +Glenohumeral Rotational Exercise Group
  Arms: Scapula Retraction +Glenohumeral Rotational Exercise Group

SUMMARY:
Abnormal reduction of the AHD has been considered as one of the possible mechanisms in the aetiology of subacromial pain syndrome. Maintenance of the AHD is crucial for prevention and rehabilitation of rotator cuff related disorders.

The development of a rehabilitation treatment plan is based in part on the assessment of scapular motion and muscle deficits in patients with shoulder pain. Rehabilitation should be based on the identified impairments.

The aim of this study is to investigate the effect of utilizing scapula retraction exercises with or without glenohumeral rotational exercises at gradual shoulder elevation angles into a scapular stabilization program on functionality, pain and AHD in patients with SPS and compare with health population.

DETAILED DESCRIPTION:
Coordinated motion between the humerus and scapula is required for pain-free arm movement. Rotator cuff and scapulothoracic muscles dynamically control the subacromial space or acromiohumeral distance (AHD).Scapulothoracic muscles need to provide stability and control in a synchronized fashion to facilitate normal scapulohumeral movement. Scapular upward rotation and posterior tilt is essential to maintain the AHD.Therefore, the force couple function of the rotator cuff muscles play an critical role in opposing the superior migration force that is generated by deltoid muscle and, to maintenance the subacromial space.

Abnormal reduction of the AHD has been considered as one of the possible mechanisms in the aetiology of subacromial impingement syndrome. Maintenance of the AHD is crucial for prevention and rehabilitation of rotator cuff related disorders.

The development of a rehabilitation treatment plan is based in part on the assessment of scapular motion and muscle deficits in patients with shoulder pain. Rehabilitation should be based on the identified impairments.

he aim of this study is to investigate the effect of utilizing scapula retraction exercises with or without glenohumeral rotational exercises at gradual shoulder elevation angles into a scapular stabilization program on functionality, pain and AHD in patients with SPS and compare with health population.

ELIGIBILITY:
Inclusion Criteria:

* painful arc of movement during flexion or abduction;
* positive Neer or Kennedy-Hawkins impingement signs
* pain on resisted lateral rotation, abduction or empty can test.

Exclusion Criteria:

* previous shoulder surgery;
* shoulder pain reproduced by neck movement;
* clinical signs of full-thickness RC tears; or
* shoulder capsulitis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Functional Level | ffrom baseline to twelve week after treatment sessions
  Functional level will be assessed by using Shoulder Pain and Disability Index (SPADİ). All assessment will be recorded at baseline, at the end of the 12-week treatment sessions and 6-month follow-up.

OTHER OUTCOMES:
pain assessment | from baseline to 6-month follow up
  pain intensity will de assessed by using Visual Analog Scale at rest, activity and at night. All assessment will be recorded at baseline, at the end of the 12-week treatment sessions and 6-month follow-up.
Acromiohumeral Distance Measurement | from baseline to 6-month follow up
  Acromiohumeral Distance will be measured by 0°, 30°, 45°, 60° and 90° of shoulder abduction positions. All assessment will be recorded at baseline, at the end of the 12-week treatment sessions and 6-month follow-up.
Patient Satisfaction | at 12 week and 6-month follow ups
  Patient Satisfaction will be assessed by simple questions consisting of self- recovery rate and patients expectation

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Health Sciences, Dept. of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We will share IPD when we recruiting the patients